CLINICAL TRIAL: NCT05519267
Title: A Randomised Trial of Mindfulness-based Social Work and Self-Care Among Social Workers
Brief Title: Mindfulness-based Social Work and Self-Care (MBSWSC)
Acronym: MBSWSC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Karen McGuigan, Dr, Queen's University, Belfast
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: REF 204_2021
Record Dates: First submitted 2022-08-18; First posted 2022-08-29 (Actual); Last update posted 2022-08-29 (Actual); Status verified 2022-08

CONDITIONS: Stress; Burnout, Professional; Anxiety; Depression; Wellbeing
MeSH Terms: conditions — Burnout, Professional; Anxiety Disorders; Depression | interventions — Self Care; Mindfulness

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBSWSC programme (Experimental): The Experimental group will take part in the Mindfulness Based Social Work and Self Care (MBSWSC) programme (6 sessions). MBSWSC will be facilitated by two accredited mindfulness practitioners, who are also qualified social workers. Sessions will be supplemented by brief homework activities.
  Interventions: Behavioral: MBSWSC
- MBSC Programme (Active Comparator): The Active comparator group will take part in the Mindfulness and Self-compassion (MBSC) programme (3 sessions). MBSC will be facilitated by two accredited mindfulness practitioners, who are also qualified social workers. Sessions will be supplemented by brief homework activities.
  Interventions: Behavioral: MBSC

INTERVENTIONS:
Behavioral: MBSWSC — MBSWSC is a unique mindfulness-based programme for social work and self-care which has been specifically developed for online delivery. The MBSWSC programme is embedded within key cognitive and emotion regulation, and stress coping theory (Maddock et al. 2019a). This programme combines mindfulness practices with psychoeducation with the aim of allowing participants to reduce any negative thinking about the past and future by learning skills that will allow them to focus on the present. It will also focus on how to effectively apply these newly acquired mindfulness skills in social work practice. The MBSWSC programme comprises 6x1.5 hour sessions, delivered weekly, over a 6 week period. Homework, in the form of mindfulness practices, is given each week. This will take approximately 20-30 minutes to complete, on 6 out of 7 days, each week.
  Other Names: Mindfulness Based Social Work and Self Care
  Arms: MBSWSC programme
Behavioral: MBSC — MBSC is a modified, condensed Mindfulness Based Intervention; with a key focus on self-compassion. Key practices in this condensed programme were chosen for their relevance and utility to social workers. The MBSC programme comprises 3x1 hour sessions delivered over a 6 week period, with one session every two weeks. Homework, in the form of mindfulness practices, is given each week. This will take approximately 20-30 minutes to complete, on 6 out of 7 days, each week.
  Other Names: Mindfulness and Self Care
  Arms: MBSC Programme

SUMMARY:
Social work is a stressful occupation with social workers at high risk of job-related stress and burnout. Mindfulness has been evidenced as a promising approach for improving: recovery from stress; behavioural responses to stress; and resilience.

The main aim of the study is to examine the efficacy of a bespoke, innovative, 6-session Mindfulness Intervention for social workers (MBSWSC) in reducing social worker stress, feelings of burnout, anxiety, low mood and improving well-being. The study will also compare outcomes from the MBSWSC with a briefer, condensed 3 session mindfulness programme (MBSC).

DETAILED DESCRIPTION:
Background: Social work is a stressful occupation with social workers at high risk of burnout. It is perhaps unsurprising then that research has focused on the impact of working conditions and work-related stress in this population. COVID has seemingly intensified pressures on frontline social workers, in turn adversely impacting their health and wellbeing.

Despite awareness of the impact of social work, job-related stress, and burnout, there remains a lack of evidence on the implementation and effectiveness of interventions to mitigate these aspects and improve outcomes for social workers. A novel, innovative approach, embedded in social work practice, is needed to support and improve social worker wellbeing. Mindfulness has emerged as a promising approach evidencing success in improving: recovery, cognitive, emotional and behavioural responses to stress. Mindfulness has also been highlighted as an approach by which resilience is strengthened. Mindfulness has been found to generate positive outcomes for those working in health and social care; promoting wellbeing, increasing levels of self-care and self-compassion, reducing stress, and combating burnout. Self-care (self-compassion) has been highlighted as an important promoter of positive health effects in social work.

Although possible benefits of mindfulness for social workers have been suggested, the evidence base to support this is scant, mainly due to a scarcity of mindfulness based intervention studies aimed at social workers. Traditionally there has been a lack of evidence on the effectiveness of briefer mindfulness programmes; with recognised programmes such as MBSR and MBCT requiring significant time commitments from participants which may not be suitable for practicing professionals. In light of this; there is a clear need for high quality RCTs to add to the evidence base in this area and to inform future provision.

With this in mind, this study looked to explore the efficacy of a bespoke, innovative, 6-session Mindfulness Intervention for social workers (MBSWSC). It also served to compare the outcomes from the MBSWSC programme with a modified, condensed 3 session mindfulness programme (MBSC).

More explicitly, this RCT aims to examine the:

* Efficacy of the MBSWSC programme at improving social worker stress, feelings of burnout, anxiety, low mood and well-being (primary outcomes).
* Effectiveness of MBSWSC in improving mindfulness, attention regulation, acceptance, self-compassion, non-attachment and aversion, worry and rumination (secondary outcomes).
* Differences between MBSWSC outcomes and outcomes on the MBSC

Methods: 93 participants providing consent to participate in the study were randomised to either the experimental (MBSWSC) or active control (MBSC) groups. 62 participants completed baseline measures; with post-intervention measures completed by 47 participants.

The primary outcome of the study is the efficacy of MBSWSC on social worker stress, feelings of burnout, anxiety, low mood and well-being and secondary outcomes. The secondary outcome of the study is the differences in outcomes for MBSWSC participants and participants on the modified, condensed (briefer) MBSC. Data will be collected pre-intervention, post-intervention and at 3 month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Frontline social work practitioner; Working in Northern Ireland; Aged 18 years and over

Exclusion Criteria:

* Social workers in strategic social work roles with no contact with clients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-09-21 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-04-29 (Actual)

PRIMARY OUTCOMES:
Change in Stress measured on the Perceived Stress Scale (PSS) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Perceived Stress Scale is a 10-item, reliable and valid, measure of perceived stress. Scores on this scale can range from 0-40, with higher scores indicative of higher levels of stress
Change in Burnout measured on the Maslach Burnout Inventory (MBI) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Maslach Burnout Inventory is a 22-item, reliable and valid measure of work-related burnout. The scale comprises 3 sub scales: burnout, depersonalisation, and personal achievement. The burnout subscale was used in this study. Scores on this sub scale can range from 0-42. Scores of ≤17 on this subscale are indicative of low-level burnout; scores of 18-29 indicate moderate burnout; scores ≥30 indicate high level burnout.
Change in Anxiety measured on the Hospital Anxiety and Depression Scale (HADS-A) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Hospital Anxiety and Depression Scale is a 14-item, reliable and valid measure of anxiety and depression. 7 of the 14 items measure severity of anxiety (HADS-A). Scores on this sub scale can range from 0-21. HADS-A subscale scores of 0-7 are considered normal, whilst scores of 11 or more are classified as moderate to severe
Change in Depression measured on the Hospital Anxiety and Depression Scale (HADS) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Hospital Anxiety and Depression Scale is a 14-item reliable and valid measure of anxiety and depression. 7 of the 14 items measure severity of depression (HADS-D). Scores on this sub scale can range from 0-21. HADS-D subscale scores of 0-7 are considered normal, whilst scores of 11 or more are classified as moderate to severe
Change in Wellbeing measured on the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Warwick-Edinburgh Mental Well-being Scale is a 14 item, reliable and valid measure of mental wellbeing. Scores on this scale can range from 14-70. Lower Warwick-Edinburgh Mental Well-being Scale scores are indicative of poorer mental wellbeing

SECONDARY OUTCOMES:
Change in Mindfulness measured by on the Southampton Mindfulness Questionnaire (SMQ) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Southampton Mindfulness Questionnaire is a 16-item reliable and valid measure assessing elements of mindfulness in response to unpleasant thoughts and images. Scores on this scale range from 0-96. Higher scores on the Southampton Mindfulness Questionnaire are indicative of greater levels on mindfulness
Change in Self-compassion measured by on the Self-Compassion Scale (SCS) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Self-Compassion Scale is a 12-item reliable and valid measure of self-compassion. Scores on this scale can range from 12-60. Higher mean scores reflect higher levels of self-compassion
Change in Worry measured on the Penn State Worry Questionnaire (PSWQ) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Penn State Worry Questionnaire is a 16-item reliable and valid measure of measure of worry. Scores on this scale can range from 16-80. Higher scores on the Penn State Worry Questionnaire reflect higher levels of pervasive, intense, and uncontrollable worry
Change in Attention Regulation (Decentering) measured on the Experiences Questionnaire - Decentring (EQ-D) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  xperiences Questionnaire - Decentring is an 11-item measure of attention regulation/decentering. Scores on this scale range from 11-55. Higher scores on the xperiences Questionnaire - Decentring reflect higher levels of attention regulation
Change in Acceptance measured on the The Philadelphia Mindfulness - Acceptance Subscale (PHLMS-A) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  The Philadelphia Mindfulness - Acceptance Subscale is a 10-item reliable and valid measure of the mindfulness component of acceptance. Total scores on this sub scale range from 10-50. Lower scores on the Philadelphia Mindfulness - Acceptance subscale reflect higher levels of acceptance
Change in Non-attachment measured by the Southampton Mindfulness Questionnaire Non Attachment subscale (SMQ-LG) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Southampton Mindfulness Questionnaire Non Attachment subscale is a reliable and valid measure of Non-attachment. Scores on this sub scale range from 0-24. Higher scores on this sub scale are indicative of higher levels of non-attachment
Change in Aversion measured by the Southampton Mindfulness Questionnaire Aversion subscale (SMQ-Av) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Southampton Mindfulness Questionnaire Aversion subscale is a reliable and valid measure of Aversion. Scores on this sub scale range from 0-24. Higher scores on this sub scale are indicative of higher levels of aversion
Change in Rumination measured on the Rumination Reflection Questionnaire Rumination subscale (RRQ-R) | Pre-intervention (week 1); Post-intervention (week 8); 3-month follow-up (week 20)
  Rumination Reflection Questionnaire Rumination subscale is a 12-item measure of engagement in rumination. Scores on this scale range from 12-60. Higher scores on this scale are indicative of greater engagement in rumination

CONTACTS AND LOCATIONS:
Overall Officials: Alan Maddock, PhD, Principal Investigator — University of Dublin, Trinity College
Locations (1):
- Queen's University Belfast, Belfast, Northern Ireland, United Kingdom

REFERENCES:
- [Derived] Maddock A, McGuigan K, McCusker P. A randomised trial of Mindfulness-based Social Work and Self-Care with social workers. Curr Psychol. 2023;42(11):9170-9183. doi: 10.1007/s12144-023-04410-w. Epub 2023 Feb 25. PMID 37200547